CLINICAL TRIAL: NCT04609930
Title: Impact of Immune Checkpoint Inhibitor Therapy on Type 2 Inflammation
Acronym: ImmunEO
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0583
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-11

CONDITIONS: Patients Recieving Anti-PD-1 or Anti-PD-L1 Immunotherapies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study population: Patients in the University Hospitals of Montpellier system who have received anti-PD-1 and/or anti-PD-L1
  Interventions: Drug: Anti-PD-1 or anti-PD-L1

INTERVENTIONS:
Drug: Anti-PD-1 or anti-PD-L1 — Immunotherapy treatment via anti programmed death 1 and/or anti-programmed death ligand 1.

SUMMARY:
The primary objective of this study is to determine the impact of anti-checkpoint immunotherapy on type 2 inflammation via a retrospective analysis of % eosinophilia.

ELIGIBILITY:
Inclusion Criteria:

* Electronic patient file "DxCare" at the University Hospitals of Montpellier
* Patient has received anti-PD-1 immunotherapy --AND/OR -- anti-PD-L1 immunotherapy according to central pharmacy records

Exclusion Criteria:

* No mention of % eosinophilia in the patient file

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population corresponds to all patients within the University Hospitals of Montpellier system who received anti-PDF-1 and/or anti-PD-L1 immunotherapies.
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Change in % eosinophilia after initiation of anti-PD-1 and/or anti-PD-L1 | Before treatment (before day 0) versus after (15 days)
Change in % eosinophilia after initiation of anti-PD-1 and/or anti-PD-L1 | Before treatment (before day 0) versus after (1 month)
Change in % eosinophilia after initiation of anti-PD-1 and/or anti-PD-L1 | Before treatment (before day 0) versus after (3 months)
Change in % eosinophilia after initiation of anti-PD-1 and/or anti-PD-L1 | Before treatment (before day 0) versus after (6 months)
Change in % eosinophilia after initiation of anti-PD-1 and/or anti-PD-L1 | Before treatment (before day 0) versus after (12 months)

SECONDARY OUTCOMES:
Indication leading to anti-PD-1 and/or anti-PD-L1 immunotherapies | Day 0
  Name of pathology
Age (years) | Day 0
Sex (male/female) | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Charriot, MD, Study Director — University Hospital, Montpellier
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No